CLINICAL TRIAL: NCT02394925
Title: Acceptance & Tolerance Study of Multifocal Contact Lenses by Functional Emmetropes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johnson & Johnson Vision Care, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CR-5672
Record Dates: First submitted 2015-03-16; First posted 2015-03-20 (Estimated); Results first posted 2017-05-15 (Actual); Last update posted 2018-06-19 (Actual); Status verified 2017-04

CONDITIONS: Vision Correction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Multifocal Test Contact Lens (Experimental): Subjects will wear the test lenses at least six hours per day, at least five days per week
  Interventions: Device: Multifocal Test Contact lens

INTERVENTIONS:
Device: Multifocal Test Contact lens — Used in a daily wear modality
  Other Names: etafilcon A

SUMMARY:
The primary objective of this study is to determine the retention rate over a two month period of vision correction in emmetropic, presbyopes fitted with multifocal contact lenses.

ELIGIBILITY:
Inclusion Criteria:

1. The subject must read, understand and sign the Statement of Informed Consent and receive a fully executed copy of the form.
2. The subject must appear able and willing to adhere to the instructions set forth in this clinical protocol.
3. The subject must be between 40 and 70 years of age.
4. The subject's vertex corrected spherical equivalent distance refraction must be in the range of -1.00 to +2.00 in each eye.
5. The subject's refractive cylinder must be less than or equal to -0.75 D in each eye.
6. The subject's ADD power must be in the range of +0.75 D to +2.50.
7. The subject must have best corrected visual acuity of 20/25 or better in each eye.

Exclusion Criteria:

1. Currently pregnant or lactating (subjects who become pregnant during the study will be discontinued).
2. Any ocular or systemic allergies that contraindicate contact lens wear.
3. Any ocular or systemic disease, autoimmune disease, or use of medication, that contraindicates contact lens wear.
4. Any ocular abnormality that may interfere with contact lens wear.
5. Use of any ocular medication, with the exception of rewetting drops.
6. Any previous intraocular surgery (e.g. radial keratotomy, PRK, LASIK, etc.).
7. Any grade 3 or greater slit lamp findings (e.g. edema, corneal neovascularization, corneal staining, tarsal abnormalities, conjunctival injection) which may contraindicate contact lens wear.
8. History of herpetic keratitis.
9. Any ocular infection or inflammation.
10. Any corneal distortion or irregular cornea.
11. History of binocular vision abnormality or strabismus.
12. Any infectious disease (e.g. hepatitis, tuberculosis) or a contagious immunosuppressive disease (e.g. HIV).
13. History of diabetes.
14. Current or previous history of being prescribed a correction for distance vision.
15. Current or previous history of contact lens wear.
16. Participation in any contact lens or lens care product clinical trial within 30 days prior to study enrollment.

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 113 (Actual)
Dates: Start 2015-01-01 (Actual); Primary Completion 2015-09-01 (Actual); Study Completion 2015-09-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (2):
- Tallahassee Eye Center, Pensacola, Florida, United States
- Ocular Technology Group-International, London, United Kingdom

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 113 enrolled into this study. Of the enrolled, 5 subjects did not meet the eligibility criteria and 108 subjects were dispensed the study lens. Of the dispensed subjects 79 completed the study while 29 subjects were discontinued.
Groups:
- Etafilcon -PVP (Multi-focal): All subjects in the study wore the test lens etafilcon- PVP (Multi-focal) throughout the entire duration of the study.
Period: Overall Study
Arm/Group | Etafilcon -PVP (Multi-focal)
Started | 108
Completed | 79
Not Completed | 29
Not completed — Adverse Event | 1
Not completed — Lens Discomfort | 3
Not completed — Lens handling difficulities | 5
Not completed — Lost to Follow-up | 9
Not completed — Protocol Violation | 5
Not completed — No longer meet eligibility criteria | 1
Not completed — Unsatisfactory Visual Response | 5

BASELINE CHARACTERISTICS:
Population: All subjects that were dispensed the study lens.
Groups:
- Dispensed Subjects: All subjects in that were dispensed the study lens.
Arm/Group | Dispensed Subjects
Number analyzed (Participants) | 108
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.9 (6.13)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 61
  Male | 47
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 31
  White | 73
  More than one race | 0
  Unknown or Not Reported | 3
Region of Enrollment [Number; unit: participants]
  United States | 46
  United Kingdom | 62

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Successful Contact Lens Wearers
Description: Proportion of Successful contact lens wearers is based on a subject's responses to two questionnaire items, "Overall Quality of Vision" and "Overall Comfort". Each item uses a 6 response like-rt scale (0= Not Applicable, 1=Excellent, 2=Very Good, 3=Good, 4=Fair and 5=Poor). The data from each item was dichotomized into two groups. If a subject responded "Excellent", "Very Good" or "Good" then the response=1, otherwise the response=0. The proportion of subjects with response=1 was reported as the proportion of successful contact lens wearers.
Time Frame: 2 months post wear
Population: Subjects that completed all study visits without a major protocol deviation.
Measure: Number; unit: Proportion of Subjects
Arm/Group | Etafilcon -PVP (Multi-focal)
Number analyzed (Participants) | 78
Proportion of Subjects | 0.71

ADVERSE EVENTS:
Time Frame: Throughout the duration of the study. Approximately 2-months per subject.
Arm/Group | Etafilcon -PVP (Multi-focal)
Serious Adverse Events (participants affected / at risk) | 0/108
Other Adverse Events (participants affected / at risk) | 0/108

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days